CLINICAL TRIAL: NCT07186075
Title: The Effect of Adolescent Mental Health Literacy Education on Mental Health Literacy and Phubbing Levels in Adolescent
Status: Completed | Type: Observational
Sponsor: Merve Akman (Other)
Collaborators: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Sponsor-Investigator, Merve Akman, specialist nurse, Zonguldak Bulent Ecevit University
Organization: Zonguldak Bulent Ecevit University (Other)
Other Study IDs: 464489
Record Dates: First submitted 2025-09-11; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Literacy
Keywords: Phubbing; Mental health literacy; Adolescent

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intervention group: 18 students
  Interventions: Behavioral: Phubbing and Mental Health Literacy Education for Adolescents
- control group: 18 students
  Interventions: Behavioral: no training was provided

INTERVENTIONS:
Behavioral: Phubbing and Mental Health Literacy Education for Adolescents — Phubbing and Mental Health Literacy Education for Adolescents
  Groups: intervention group
Behavioral: no training was provided — no training was provided
  Groups: control group

SUMMARY:
The aim of this research, conducted with an experimental model, is to determine the effectiveness of "Phubbing and Mental Health Literacy Education for Adolescents" on phubbing and mental health literacy levels in high school students. The research was conducted in two Anatolian high schools in Zonguldak. The study sample consisted of 36 adolescents between the ages of 15 and 17 with high levels of phubbing and low levels of mental health literacy (intervention group= 18, control group= 18). Data were collected using the "Personal Information Form," the "General Phubbing Scale," and the "Adolescent Mental Health Literacy Scale" in three stages: pre-test, post-test, and follow-up test. "Phubbing and Mental Health Literacy Education for Adolescents" was applied to the intervention group.

H1: Phubbing and mental health literacy education for adolescents has an effect on reducing the level of phubbing.

H2: Phubbing and mental health literacy education for adolescents has an effect on increasing the level of mental health literacy.

ELIGIBILITY:
Inclusion Criteria:

Being a volunteer

* Being in the 10th or 11th grade
* The adolescent must have a smartphone
* The adolescent must have a high phubbing scale score and a low adolescent mental health literacy scale score
* The adolescent must not have any auditory, visual or learning disabilities
* Being able to speak and understand Turkish

Exclusion Criteria:

Not volunteering

* Being in the 9th or 12th grade
* Not having a smartphone
* Having a low phubbing scale score and a high adolescent mental health literacy scale score
* Having any learning disabilities
* Not being able to speak and understand Turkish

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The research was conducted in two Anatolian high schools in Zonguldak. The study sample consisted of 36 adolescents between the ages of 15 and 17 with high levels of phubbing and low levels of mental health literacy (intervention group= 18, control group= 18).
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
The Adolescent Mental Health Literacy Scale | up to six weeks after the end of the training.
  The effectiveness of mental health literacy training in adolescents was evaluated. The "Adolescent Mental Health Literacy Scale" was used to measure students' mental health literacy levels. Students' mental health literacy data were measured using a pretest, posttest, and follow-up test.
The General Phubbing Scale | up to six weeks after the end of the training.
  The effectiveness of phubbing and mental health literacy training in adolescents was evaluated. The "General Phubbing Scale" was used to measure students' phubbing levels. Students' phubbing data were measured using a pretest, posttest, and follow-up test.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol